CLINICAL TRIAL: NCT05613101
Title: Comparison of the Effects of Ultrasound-Guided Erector Spinae Plane Block and Adductor Canal Block on Postoperative Pain, Opioid Consumption and Quadriceps Muscle Strength in Total Knee Arthroplasty Surgery
Brief Title: ESPB and ACB in Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, İnal Bensu Arıoglu, Medical Doctor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulMUG
Record Dates: First submitted 2022-10-06; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Post Operative Pain
Keywords: Erector Spinae Plane Block; Adductor Canal Block; Total Knee Arthroplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Erector Plane Block Adductor Canal Block
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): Erector Spina Plane Block was performed to the patients after coplition of total knee arthroplasty operation for postopetaive pain.
  Interventions: Procedure: Erector Spinae Plane Block
- Adductor Canal Block (Active Comparator): Adductor Canal Block was performed to the patients after coplition of total knee arthroplasty operation for postopetaive pain.
  Interventions: Procedure: Adductor Canal Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — After the necessary asepsis and antisepsis procedures, the linear ultrasound probe was placed parasagittally 2-3 cm lateral to the spinous process at the L3 or L4 level and the transverse process was visualized. The peripheral block needle (85 mm B Braun Stimuplex A) was advanced in plane up to the transverse process and 10 ml 0.5% bupivacaine hydrochloride 10 ml 0.9% isotonic NaCl mixture was applied on the erector spina muscle.
  Arms: Erector Spinae Plane Block
Procedure: Adductor Canal Block — After the necessary asepsis and antisepsis procedures, the linear ultrasound probe was placed in the middle between the medial condyle and the SIAS, and the superficial femoral artery (FSA) was visualized under the sartorius muscle. By following the FSA distally, the point where the sartorius muscle crosses the adductor magnus muscle, which is the beginning of the adductor canal, was found and the saphenous nerve was visualized hyperechoic in the anterolateral aspect of the FSA. 20 cc 0.5% bupivacaine hydrochloride was applied
  Arms: Adductor Canal Block

SUMMARY:
Total knee arthroplasty surgery is preferred in the treatment of osteoarthritis and causes severe postoperative pain. In this study, we aimed to investigate the effects of lumbar erector spina plan block and adductor canal block on postoperative pain and quadriceps muscle strength in patients who underwent total knee arthroplasty with spinal anesthesia.

DETAILED DESCRIPTION:
In a prospective, randomized study; Medeniyet University Faculty of Medicine Göztepe Prof. Dr. Forty patients who underwent total knee arthroplasty surgery at Süleyman Yalçın City Hospital were divided into two groups. After the surgery was completed, erector spina plane block was applied to Group E (n=20) patients with 20 ml of 0.25% bupivacaine from the operated side L3-L4 level, while in Group A (n=20) patients, in the area where the sartorius muscle crosses the adductor magnus muscle, it was lateral to the superficial femoral artery. Adductor canal block was applied to the adductor canal with 20 ml of 0.5% bupivacaine. All patients were administered 1 gr paracetamol and 75 mg diclofenac sodium when their pain started in the orthopedic ward. Numerical pain score and quadriceps muscle strength were evaluated during the 48-hour follow-up of the patients. When the pain score was 4 and above, 50 mg pethidine hydrochloride was administered.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent total knee arthroplasty surgery
* ASA I-III patients

Exclusion Criteria:

* Patients with coagulopathy
* Patients history with local anesthetic allergy or toxicity
* Patients with long hospital stay
* Patients with advanced organ failure
* Mental retarded patients
* Presence of infection at the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain 30 minute | 30. min.
  Visual anolog score (1-10)
Postoperative pain 1. hour | 1. hour
  Visual anolog score (1-10)
Postoperative pain 2. hour | 2. hour
  Visual anolog score (1-10)
Postoperative pain 6. hour | 6. hour
  Visual anolog score (1-10)
Postoperative pain 12. hour | 12. hour
  Visual anolog score (1-10)
Postoperative pain 24. hour | 24. hour
  Visual anolog score (1-10)
Postoperative pain 36. hour | 36. hour
  Visual anolog score (1-10)
Postoperative pain 48. hour | 48. hour
  Visual anolog score (1-10)

SECONDARY OUTCOMES:
Opioid consuption 30. min. | 30. min.
  Petidine (mg)
Opioid consuption 1. hour | 1. hour
  Petidine (mg)
Opioid consuption 2. hour | 2. hour
  Petidine (mg)
Opioid consuption 6. hour | 6. hour
  Petidine (mg)
Opioid consuption 12. hour | 12. hour
  Petidine (mg)
Opioid consuption 24. hour | 24. hour
  Petidine (mg)
Opioid consuption 36. hour | 36. hour
  Petidine (mg)
Opioid consuption 48. hour | 48. hour
  Petidine (mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Goztepe Suleyman Yalcın City Hospital, Istanbul, Turkey (Türkiye)